CLINICAL TRIAL: NCT02653196
Title: A Multi-Institutional Pilot Study of Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Malignant Neuro-Epithelial and Other Solid Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The Principal Investigator left the institution.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Children's Hospital Los Angeles (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Kris M. Mahadeo, Assistant Professor, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-3856
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-06

CONDITIONS: Neuroepithelial Tumor; Solid Tumor; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Neoplasms, Neuroepithelial | interventions — Fibroblast Growth Factor 7; Alemtuzumab; Thiotepa; Etoposide; fludarabine; fludarabine phosphate; Melphalan; Tacrolimus; Cyclosporine; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Hematopoietic Stem Cell Transplant (Experimental): Matched Unrelated Donor HSCT (minimum 9/10 human leukocyte antigen [HLA] match) OR Matched Related Donor HSCT (10/10 HLA match). Conditioning regimen begins 12 days prior to stem cell infusion and includes the following drugs:
  Keratinocyte Growth Factor Alemtuzumab Thiotepa Etoposide Melphalan Fludarabine Tacrolimus (Cyclosporine A may be substituted for Tacrolimus) Mycophenolate mofetil
  Interventions: Procedure: Allogeneic hematopoietic stem cell transplant following thiotepa-based marrow ablative chemotherapy; Drug: Keratinocyte Growth Factor; Drug: Alemtuzumab; Drug: Thiotepa; Drug: Etoposide; Drug: Fludarabine; Drug: Melphalan; Drug: Tacrolimus; Drug: Cyclosporine A; Drug: Mycophenolate mofetil

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem cell transplant following thiotepa-based marrow ablative chemotherapy — Allogeneic hematopoietic stem cell transplant (HSCT) following thiotepa-based marrow ablative chemotherapy (MAC) for children with high-grade and/or recurrent neuro-epithelial and other solid tumors.
Drug: Keratinocyte Growth Factor — KGF 60 mcg/kg IV: 6 doses
  Other Names: KGF; Kepivance; Palifermin
Drug: Alemtuzumab — Alemtuzumab 12 mg/m2 IV: 2 doses (not given if matched related donor is 10/10 HLA matched sibling donor)
  Other Names: Campath; Campath 1H
Drug: Thiotepa — Thiotepa 300 mg/m2 IV: 3 doses
Drug: Etoposide — Etoposide 100 mg/m2 IV: 3 doses
  Other Names: VP-16
Drug: Fludarabine — Fludarabine 30 mg/m2 IV: 3 doses
  Other Names: FLUDARA
Drug: Melphalan — Melphalan 70 mg/m2 IV: Day 2 doses
Drug: Tacrolimus — Tacrolimus 0.05 mg/kg/day IV (Cyclosporine may be substituted for Tacrolimus): Start Day -2, begin taper on Day +100, discontinue on Day +180
Drug: Cyclosporine A — Cyclosporine A dosed as follows: Age ≤ 6 years: 6 mg/kg/day IV in divided doses (e.g. 2 mg/kg every 8 hours) OR Age > 6 years: 3 mg/kg/day IV in divided doses (1.5 mg/kg every 12 hours): Start Day -2, begin taper on Day +100, discontinue on Day +180
  Other Names: Cyclosporine; CYA; CSA; Sandimmune; Neoral; Gengraf
Drug: Mycophenolate mofetil — Mycophenolate mofetil 15 mg/kg every 8 hours oral or IV: Start Day 0 (4-6 hours post stem cell infusion) to Day +40, then taper weekly until discontinuation on Day +90
  Other Names: MMF; Cellcept; Myfortic

SUMMARY:
There is currently no standard treatment for patients with neuro-epithelial (brain) or other solid tumors in another part of the body who do not have adequate suitable autologous hematopoietic progenitor cells available and/or whose disease has relapsed after standard treatment. Allogeneic Hematopoietic Progenitor Cell Transplant may be a consideration for treatment of patients with recurrent chemo-responsive malignant (high grade) neuro-epithelial and other solid tumors or those who do not have suitable autologous hematopoietic progenitor cell availability. The procedure in which your own blood stem cells are transplanted to you is called an autologous (from your own) progenitor cell transplant and when cells from a matched donor are transfused is called an allogeneic progenitor cell transplant. The study is being conducted to evaluate the safety and effectiveness of a combination of drugs followed by an allogeneic hematopoietic progenitor cell transplant (HPCT). This treatment regimen is experimental in that although the individual drugs are commonly used to treat your disease, the specific combination used in this protocol followed by the transplant is experimental.

DETAILED DESCRIPTION:
This is a multi-institutional Pilot clinical trial of hematopoietic stem cell transplantation (HSCT) for (i) patients with recurrent chemo-responsive malignant (high-grade) neuro-epithelial and other solid tumors which are recurrent following HSCT or (ii) for said patients without autologous hematopoietic progenitor cell availability. The stem cells will be derived from a 1) matched related donor or 2) matched unrelated donor (MUD).

This is a pilot study of a novel HSCT protocol for patients with high-grade and/or recurrent neuro-epithelial and other solid tumors. To determine the feasibility of allogeneic HSCT following thiotepa-based marrow ablative chemotherapy (MAC) for children with high-grade and/or recurrent neuro-epithelial and other solid tumors. The primary end-point for this study is to determine progression-free survival (PFS) at six months post-HSCT. Secondary end-points include: (a) overall survival (OS) at one year (b) transplant related mortality (TRM) at Day +100 (c) engraftment (d) regimen related toxicity: the frequency and severity of acute and chronic graft-versus-host disease (GVHD), sinusoidal obstructive syndrome and infections will be assessed (e) time to immune reconstitution following HSCT. Exploratory Aims include: 1) To assess the feasibility of the Taqman® Low Density Arrays (TLDA) assay as a technology for MRD detection among a subset of patients with high-grade and/or recurrent neuro-epithelial and other solid tumors. Minimal residual disease (MRD) (when applicable) in bone marrow pre- and post-HSCT, will be assessed using TLDA. Currently, for solid malignancies there is no routinely established method to detect minimal residual disease, the first indicator of therapy failure and/or recurrence of disease. 2) In an effort to minimize morbidity related to graft-versus-host disease, alemtuzumab forms an important component of the proposed MAC regimen for recipients of unrelated or related mismatched allogeneic grafts. As an exploratory aim, an alemtuzumab assay will be performed at specified intervals to explore time to drug clearance. This may provide important information regarding lymphodepletion for future trials regarding immunotherapy administered during recovery from HSCT therapy.

The main advantages of the proposed approach will: 1) Overcome the challenges in bone morrow/peripheral blood stem cell (PBSC) collection in patients heavily pre-treated and/or bone/bone marrow infiltration with tumor. 2) Eliminate the risk of graft contamination with tumor cells, and 3) Graft-versus-tumor effect (GVT) to eliminate residual disease after conditioning chemotherapy. The use of allografting with the proposed regimen combines the benefits of high dose chemotherapy and an immune approach to disease therapy.

ELIGIBILITY:
Inclusion Criteria:

* Malignant (high-grade) neuro-epithelial and other solid tumors
* Patients have to be in at least, a chemo-responsive disease status defined as; any disease regression to chemotherapy when compared to its pre-treatment evaluation
* Patients with recurrent (or refractory) chemo-responsive disease or without suitable autologous hematopoietic progenitor cell availability
* Creatinine clearance or glomerular filtration rate (GFR) ≥50 ml/min/1.73m2, and not requiring dialysis
* Diffusing capacity of lung for carbon monoxide, or DLCO, (corrected for hemoglobin) ≥ 50% predicted. If unable to perform pulmonary function tests, then oxygen (O2) saturation ≥ 92% in room air
* Bilirubin ≤3x upper limit of normal (ULN) and alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 5x for age (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome)

Exclusion Criteria:

* Lack of histocompatible suitable related or unrelated donor/ graft source
* End-organ failure that precludes the ability to tolerate the transplant procedure, including conditioning
* Renal failure requiring dialysis
* Congenital heart disease resulting in congestive heart failure
* Ventilatory failure
* HIV infection
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication yet clinical symptoms progress); stable, controlled disease with treatment is not an exclusion criteria
* Female of reproductive potential who is pregnant, planning to become pregnant during the study, or is nursing a child

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | Six months post-transplant

SECONDARY OUTCOMES:
Overall Survival | One year post-transplant
Transplant Related Mortality | Day +100 post-transplant
Engraftment | Within 100 days post-transplant
Regimen Related Toxicity | Within one year post-transplant
  Frequency and severity of acute and chronic graft-versus-host disease
Time to Immune Reconstitution | Within one year post-transplant

OTHER OUTCOMES:
Feasibility of Taqman® Low Density Arrays (TLDA) | Prior to stem cell infusion to one year post-transplant, at specified intervals.
  Use of TLDA assay as a technology for MRD detection among a subset of patients with high-grade and/or recurrent neuro-epithelial and other solid tumors.
Alemtuzumab Assay | Ten days prior to stem cell infusion to 28 days post-transplant, at specified intervals
  The Alemtuzumab assay will explore time to drug clearance. This may provide important information regarding lymphodepletion for future trials regarding immunotherapy administered during recovery from HSCT therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kris M Mahadeo, MD,MPH, Principal Investigator — The Children's Hospital at Montefiore
Locations (1):
- The Children's Hospital at Montefiore, The Bronx, New York, United States

REFERENCES:
- [Background] Smith MA, Seibel NL, Altekruse SF, Ries LA, Melbert DL, O'Leary M, Smith FO, Reaman GH. Outcomes for children and adolescents with cancer: challenges for the twenty-first century. J Clin Oncol. 2010 May 20;28(15):2625-34. doi: 10.1200/JCO.2009.27.0421. Epub 2010 Apr 19. PMID 20404250
- [Background] Chow KH, Gottschalk S. Cellular immunotherapy for high-grade glioma. Immunotherapy. 2011 Mar;3(3):423-34. doi: 10.2217/imt.10.110. PMID 21395383
- [Background] Daniels BP, Cruz-Orengo L, Pasieka TJ, Couraud PO, Romero IA, Weksler B, Cooper JA, Doering TL, Klein RS. Immortalized human cerebral microvascular endothelial cells maintain the properties of primary cells in an in vitro model of immune migration across the blood brain barrier. J Neurosci Methods. 2013 Jan 15;212(1):173-9. doi: 10.1016/j.jneumeth.2012.10.001. Epub 2012 Oct 13. PMID 23068604
- [Background] Mitchell DA, Fecci PE, Sampson JH. Immunotherapy of malignant brain tumors. Immunol Rev. 2008 Apr;222:70-100. doi: 10.1111/j.1600-065X.2008.00603.x. PMID 18363995
- [Background] Packer RJ, Gajjar A, Vezina G, Rorke-Adams L, Burger PC, Robertson PL, Bayer L, LaFond D, Donahue BR, Marymont MH, Muraszko K, Langston J, Sposto R. Phase III study of craniospinal radiation therapy followed by adjuvant chemotherapy for newly diagnosed average-risk medulloblastoma. J Clin Oncol. 2006 Sep 1;24(25):4202-8. doi: 10.1200/JCO.2006.06.4980. PMID 16943538
- [Background] Finlay JL, Goldman S, Wong MC, Cairo M, Garvin J, August C, Cohen BH, Stanley P, Zimmerman RA, Bostrom B, Geyer JR, Harris RE, Sanders J, Yates AJ, Boyett JM, Packer RJ. Pilot study of high-dose thiotepa and etoposide with autologous bone marrow rescue in children and young adults with recurrent CNS tumors. The Children's Cancer Group. J Clin Oncol. 1996 Sep;14(9):2495-503. doi: 10.1200/JCO.1996.14.9.2495. PMID 8823328
- [Background] Sung KW, Yoo KH, Cho EJ, Koo HH, Lim DH, Shin HJ, Ahn SD, Ra YS, Choi ES, Ghim TT. High-dose chemotherapy and autologous stem cell rescue in children with newly diagnosed high-risk or relapsed medulloblastoma or supratentorial primitive neuroectodermal tumor. Pediatr Blood Cancer. 2007 Apr;48(4):408-15. doi: 10.1002/pbc.21064. PMID 17066462
- [Background] Ris MD, Packer R, Goldwein J, Jones-Wallace D, Boyett JM. Intellectual outcome after reduced-dose radiation therapy plus adjuvant chemotherapy for medulloblastoma: a Children's Cancer Group study. J Clin Oncol. 2001 Aug 1;19(15):3470-6. doi: 10.1200/JCO.2001.19.15.3470. PMID 11481352
- [Background] Henon PR, Butturini A, Gale RP. Blood-derived haematopoietic cell transplants: blood to blood? Lancet. 1991 Apr 20;337(8747):961-3. doi: 10.1016/0140-6736(91)91583-g. No abstract available. PMID 1678042
- [Background] Mason WP, Grovas A, Halpern S, Dunkel IJ, Garvin J, Heller G, Rosenblum M, Gardner S, Lyden D, Sands S, Puccetti D, Lindsley K, Merchant TE, O'Malley B, Bayer L, Petriccione MM, Allen J, Finlay JL. Intensive chemotherapy and bone marrow rescue for young children with newly diagnosed malignant brain tumors. J Clin Oncol. 1998 Jan;16(1):210-21. doi: 10.1200/JCO.1998.16.1.210. PMID 9440745
- [Background] Shih CS, Hale GA, Gronewold L, Tong X, Laningham FH, Gilger EA, Srivastava DK, Kun LE, Gajjar A, Fouladi M. High-dose chemotherapy with autologous stem cell rescue for children with recurrent malignant brain tumors. Cancer. 2008 Mar 15;112(6):1345-53. doi: 10.1002/cncr.23305. PMID 18224664
- [Background] Gururangan S, Krauser J, Watral MA, Driscoll T, Larrier N, Reardon DA, Rich JN, Quinn JA, Vredenburgh JJ, Desjardins A, McLendon RE, Fuchs H, Kurtzberg J, Friedman HS. Efficacy of high-dose chemotherapy or standard salvage therapy in patients with recurrent medulloblastoma. Neuro Oncol. 2008 Oct;10(5):745-51. doi: 10.1215/15228517-2008-044. Epub 2008 Aug 28. PMID 18755919
- [Background] Butturini AM, Jacob M, Aguajo J, Vander-Walde NA, Villablanca J, Jubran R, Erdreich-Epstein A, Marachelian A, Dhall G, Finlay JL. High-dose chemotherapy and autologous hematopoietic progenitor cell rescue in children with recurrent medulloblastoma and supratentorial primitive neuroectodermal tumors: the impact of prior radiotherapy on outcome. Cancer. 2009 Jul 1;115(13):2956-63. doi: 10.1002/cncr.24341. PMID 19402050
- [Background] Lundberg JH, Weissman DE, Beatty PA, Ash RC. Treatment of recurrent metastatic medulloblastoma with intensive chemotherapy and allogeneic bone marrow transplantation. J Neurooncol. 1992 Jun;13(2):151-5. doi: 10.1007/BF00172764. PMID 1432032
- [Background] Secondino S, Pedrazzoli P, Schiavetto I, Basilico V, Bramerio E, Massimino M, Gambacorta M, Siena S. Antitumor effect of allogeneic hematopoietic SCT in metastatic medulloblastoma. Bone Marrow Transplant. 2008 Jul;42(2):131-3. doi: 10.1038/bmt.2008.86. Epub 2008 Mar 31. No abstract available. PMID 18372908
- [Background] Takada S, Ito K, Sakura T, Hatsumi N, Sato M, Saito T, Shiozaki H, Matsushima T, Miyawaki S. Three AML patients with existing or pre-existing intracerebral granulocytic sarcomas who were successfully treated with allogeneic bone marrow transplantations. Bone Marrow Transplant. 1999 Apr;23(7):731-4. doi: 10.1038/sj.bmt.1701635. PMID 10218852
- [Background] Kasow KA, Handgretinger R, Krasin MJ, Pappo AS, Leung W. Possible allogeneic graft-versus-tumor effect in childhood melanoma. J Pediatr Hematol Oncol. 2003 Dec;25(12):982-6. doi: 10.1097/00043426-200312000-00016. PMID 14663285
- [Background] Ueno NT, Cheng YC, Rondon G, Tannir NM, Gajewski JL, Couriel DR, Hosing C, de Lima MJ, Anderlini P, Khouri IF, Booser DJ, Hortobagyi GN, Pagliaro LC, Jonasch E, Giralt SA, Champlin RE. Rapid induction of complete donor chimerism by the use of a reduced-intensity conditioning regimen composed of fludarabine and melphalan in allogeneic stem cell transplantation for metastatic solid tumors. Blood. 2003 Nov 15;102(10):3829-36. doi: 10.1182/blood-2003-04-1022. Epub 2003 Jul 24. PMID 12881308
- [Background] Ruggeri L, Capanni M, Urbani E, Perruccio K, Shlomchik WD, Tosti A, Posati S, Rogaia D, Frassoni F, Aversa F, Martelli MF, Velardi A. Effectiveness of donor natural killer cell alloreactivity in mismatched hematopoietic transplants. Science. 2002 Mar 15;295(5562):2097-100. doi: 10.1126/science.1068440. PMID 11896281
- [Background] Venstrom JM, Zheng J, Noor N, Danis KE, Yeh AW, Cheung IY, Dupont B, O'Reilly RJ, Cheung NK, Hsu KC. KIR and HLA genotypes are associated with disease progression and survival following autologous hematopoietic stem cell transplantation for high-risk neuroblastoma. Clin Cancer Res. 2009 Dec 1;15(23):7330-4. doi: 10.1158/1078-0432.CCR-09-1720. Epub 2009 Nov 24. PMID 19934297
- [Background] Aoyama Y, Yamamura R, Shima E, Nakamae H, Makita K, Kho G, Ohta K, Yamane T, Takubo T, Hino M. Successful treatment with reduced-intensity stem cell transplantation in a case of relapsed refractory central nervous system lymphoma. Ann Hematol. 2003 Jun;82(6):371-3. doi: 10.1007/s00277-003-0651-z. Epub 2003 Apr 29. PMID 12719887
- [Background] Varadi G, Or R, Kapelushnik J, Naparstek E, Nagler A, Brautbar C, Amar A, Kirschbaum M, Samuel S, Slavin S, Siegal T. Graft-versus-lymphoma effect after allogeneic peripheral blood stem cell transplantation for primary central nervous system lymphoma. Leuk Lymphoma. 1999 Jun;34(1-2):185-90. doi: 10.3109/10428199909083396. PMID 10350348
- [Background] Abdel-Azim H, Kapoor N, Mahadeo KM, Finlay JL. Graft versus tumor effect in the brain of a child with recurrent metastatic medulloblastoma. Pediatr Blood Cancer. 2015 Sep;62(9):1667-9. doi: 10.1002/pbc.25525. Epub 2015 Apr 20. PMID 25894457
- [Background] Ellman L, Katz DH, Green I, Paul WE, Benacerraf B. Mechanisms involved in the antileukemic effect of immunocompetent allogeneic lymphoid cell transfer. Cancer Res. 1972 Jan;32(1):141-8. No abstract available. PMID 4400015
- [Background] Symons HJ, Levy MY, Wang J, Zhou X, Zhou G, Cohen SE, Luznik L, Levitsky HI, Fuchs EJ. The allogeneic effect revisited: exogenous help for endogenous, tumor-specific T cells. Biol Blood Marrow Transplant. 2008 May;14(5):499-509. doi: 10.1016/j.bbmt.2008.02.013. PMID 18410892
- [Background] Maine GN, Mule JJ. Making room for T cells. J Clin Invest. 2002 Jul;110(2):157-9. doi: 10.1172/JCI16166. No abstract available. PMID 12122106
- [Background] Ahmed N, Ratnayake M, Savoldo B, Perlaky L, Dotti G, Wels WS, Bhattacharjee MB, Gilbertson RJ, Shine HD, Weiss HL, Rooney CM, Heslop HE, Gottschalk S. Regression of experimental medulloblastoma following transfer of HER2-specific T cells. Cancer Res. 2007 Jun 15;67(12):5957-64. doi: 10.1158/0008-5472.CAN-06-4309. PMID 17575166
- [Background] Perez-Martinez A, de Prada Vicente I, Fernandez L, Gonzalez-Vicent M, Valentin J, Martin R, Maxwell H, Sevilla J, Vicario JL, Diaz MA. Natural killer cells can exert a graft-vs-tumor effect in haploidentical stem cell transplantation for pediatric solid tumors. Exp Hematol. 2012 Nov;40(11):882-891.e1. doi: 10.1016/j.exphem.2012.07.004. Epub 2012 Jul 4. PMID 22771496
- [Background] Ash S, Gigi V, Askenasy N, Fabian I, Stein J, Yaniv I. Graft versus neuroblastoma reaction is efficiently elicited by allogeneic bone marrow transplantation through cytolytic activity in the absence of GVHD. Cancer Immunol Immunother. 2009 Dec;58(12):2073-84. doi: 10.1007/s00262-009-0715-6. Epub 2009 May 13. PMID 19437016
- [Background] Lang P, Pfeiffer M, Muller I, Schumm M, Ebinger M, Koscielniak E, Feuchtinger T, Foll J, Martin D, Handgretinger R. Haploidentical stem cell transplantation in patients with pediatric solid tumors: preliminary results of a pilot study and analysis of graft versus tumor effects. Klin Padiatr. 2006 Nov-Dec;218(6):321-6. doi: 10.1055/s-2006-942256. PMID 17080334
- [Background] Jubert C, Wall DA, Grimley M, Champagne MA, Duval M. Engraftment of unrelated cord blood after reduced-intensity conditioning regimen in children with refractory neuroblastoma: a feasibility trial. Bone Marrow Transplant. 2011 Feb;46(2):232-7. doi: 10.1038/bmt.2010.107. Epub 2010 May 3. PMID 20436519
- [Background] Koscielniak E, Gross-Wieltsch U, Treuner J, Winkler P, Klingebiel T, Lang P, Bader P, Niethammer D, Handgretinger R. Graft-versus-Ewing sarcoma effect and long-term remission induced by haploidentical stem-cell transplantation in a patient with relapse of metastatic disease. J Clin Oncol. 2005 Jan 1;23(1):242-4. doi: 10.1200/JCO.2005.05.940. No abstract available. PMID 15625381
- [Background] Burdach S, van Kaick B, Laws HJ, Ahrens S, Haase R, Korholz D, Pape H, Dunst J, Kahn T, Willers R, Engel B, Dirksen U, Kramm C, Nurnberger W, Heyll A, Ladenstein R, Gadner H, Jurgens H, Go el U. Allogeneic and autologous stem-cell transplantation in advanced Ewing tumors. An update after long-term follow-up from two centers of the European Intergroup study EICESS. Stem-Cell Transplant Programs at Dusseldorf University Medical Center, Germany and St. Anna Kinderspital, Vienna, Austria. Ann Oncol. 2000 Nov;11(11):1451-62. doi: 10.1023/a:1026539908115. PMID 11142486
- [Background] Burdach S. Treatment of advanced Ewing tumors by combined radiochemotherapy and engineered cellular transplants. Pediatr Transplant. 2004 Jun;8 Suppl 5:67-82. doi: 10.1111/j.1398-2265.2004.00186.x. PMID 15125708
- [Background] Lucas KG, Schwartz C, Kaplan J. Allogeneic stem cell transplantation in a patient with relapsed Ewing sarcoma. Pediatr Blood Cancer. 2008 Jul;51(1):142-4. doi: 10.1002/pbc.21503. PMID 18266223
- [Background] Capitini CM, Derdak J, Hughes MS, Love CP, Baird K, Mackall CL, Fry TJ. Unusual sites of extraskeletal metastases of Ewing sarcoma after allogeneic hematopoietic stem cell transplantation. J Pediatr Hematol Oncol. 2009 Feb;31(2):142-4. doi: 10.1097/MPH.0b013e31819146e5. PMID 19194203
- [Background] Hosono A, Makimoto A, Kawai A, Takaue Y. Segregated graft-versus-tumor effect between CNS and non-CNS lesions of Ewing's sarcoma family of tumors. Bone Marrow Transplant. 2008 Jun;41(12):1067-8. doi: 10.1038/bmt.2008.26. Epub 2008 Mar 10. No abstract available. PMID 18332914
- [Background] Kido A, Amano I, Honoki K, Tanaka H, Morii T, Fujii H, Yoshitani K, Tanaka Y. Allogeneic and autologous stem cell transplantation in advanced small round cell sarcomas. J Orthop Sci. 2010 Sep;15(5):690-5. doi: 10.1007/s00776-010-1504-y. Epub 2010 Oct 16. No abstract available. PMID 20953934
- [Background] Fagioli F, Berger M, Brach del Prever A, Lioji S, Aglietta M, Ferrari S, Picci P, Madon E. Regression of metastatic osteosarcoma following non-myeloablative stem cell transplantation. A case report. Haematologica. 2003 May;88(5):ECR16. PMID 12745285
- [Background] Goi K, Sugita K, Tezuka T, Sato H, Uno K, Inukai T, Hamada Y, Nakazawa S. A successful case of allogeneic bone marrow transplantation for osteosarcoma with multiple metastases of lung and bone. Bone Marrow Transplant. 2006 Jan;37(1):115-6. doi: 10.1038/sj.bmt.1705209. No abstract available. PMID 16258530
- [Background] Ohta H, Hashii Y, Yoshida H, Kusuki S, Tokimasa S, Yoneda A, Fukuzawa M, Inoue N, Hara J, Kusafuka T, Ozono K. Allogeneic hematopoietic stem cell transplantation against recurrent rhabdomyosarcoma. J Pediatr Hematol Oncol. 2011 Jan;33(1):e35-8. doi: 10.1097/MPH.0b013e3181e7ddc5. PMID 20975586
- [Background] Donker AE, Hoogerbrugge PM, Mavinkurve-Groothuis AM, van de Kar NC, Boetes C, Hulsbergen-van de Kaa CA, Groot-Loonen JJ. Metastatic rhabdomyosarcoma cured after chemotherapy and allogeneic SCT. Bone Marrow Transplant. 2009 Jan;43(2):179-80. doi: 10.1038/bmt.2008.301. Epub 2008 Sep 1. No abstract available. PMID 18762761
- [Background] Baird K, Fry TJ, Steinberg SM, Bishop MR, Fowler DH, Delbrook CP, Humphrey JL, Rager A, Richards K, Wayne AS, Mackall CL. Reduced-intensity allogeneic stem cell transplantation in children and young adults with ultrahigh-risk pediatric sarcomas. Biol Blood Marrow Transplant. 2012 May;18(5):698-707. doi: 10.1016/j.bbmt.2011.08.020. Epub 2011 Sep 5. PMID 21896345
- [Background] Childs R, Chernoff A, Contentin N, Bahceci E, Schrump D, Leitman S, Read EJ, Tisdale J, Dunbar C, Linehan WM, Young NS, Barrett AJ. Regression of metastatic renal-cell carcinoma after nonmyeloablative allogeneic peripheral-blood stem-cell transplantation. N Engl J Med. 2000 Sep 14;343(11):750-8. doi: 10.1056/NEJM200009143431101. PMID 10984562
- [Background] Scott M, Lawrance J, Dennis M. Regression of a renal cell carcinoma following allogeneic peripheral blood stem cell transplant for acute myeloid leukaemia: evidence of a graft-versus-tumour effect without significant graft-versus-host disease. Br J Haematol. 2012 Oct;159(1):1. doi: 10.1111/j.1365-2141.2012.09238.x. Epub 2012 Jul 27. No abstract available. PMID 22845006
- [Background] Baek HJ, Han DK, Hwang TJ, Bae SH, Choi YD, Kook H. Long-term graft-versus-tumor effect following reduced intensity hematopoietic stem cell transplantation in a child with metastatic renal cell carcinoma. Pediatr Blood Cancer. 2012 Sep;59(3):583-5. doi: 10.1002/pbc.24074. Epub 2012 Jan 9. PMID 22231905
- [Background] Inaba H, Handgretinger R, Furman W, Hale G, Leung W. Allogeneic graft-versus-hepatoblastoma effect. Pediatr Blood Cancer. 2006 Apr;46(4):501-5. doi: 10.1002/pbc.20404. PMID 15806543
- [Background] Pappo AS, Anderson JR, Crist WM, Wharam MD, Breitfeld PP, Hawkins D, Raney RB, Womer RB, Parham DM, Qualman SJ, Grier HE. Survival after relapse in children and adolescents with rhabdomyosarcoma: A report from the Intergroup Rhabdomyosarcoma Study Group. J Clin Oncol. 1999 Nov;17(11):3487-93. doi: 10.1200/JCO.1999.17.11.3487. PMID 10550146
- [Background] Bowers DC, Gargan L, Weprin BE, Mulne AF, Elterman RD, Munoz L, Giller CA, Winick NJ. Impact of site of tumor recurrence upon survival for children with recurrent or progressive medulloblastoma. J Neurosurg. 2007 Jul;107(1 Suppl):5-10. doi: 10.3171/PED-07/07/005. PMID 17644914